CLINICAL TRIAL: NCT06108089
Title: Novel Hypoxia Imaging for Head and Neck Cancer: Imaging Phenotype for Personalized Treatment
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Yoshimi Anzai, Principal Investigator, Professor of Radiology, University of Utah
Other Study IDs: 107380
Record Dates: First submitted 2023-10-05; First posted 2023-10-30 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer; Hypoxia; Magnetic Resonance Imaging; Cancer Neck
Keywords: hypoxia; precision medicine; imaging biomarker; prognosis
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients treated with CRT: Two hypoxia MR scans will be performed, one at pre-treatment and one at 2 weeks into CRT. Patients receive FMISO-PET/CT scans prior to the initiation of CRT.
  Interventions: Diagnostic Test: [18F]MISO-PET/CT
- patients treated with primary surgical resection.: Hypoxia MR scan and FMISO-PET/CT scan will be performed prior to the treatment (surgery). Surgical specimen of excised primary tumor will undergo IHC staining.
  Interventions: Diagnostic Test: [18F]MISO-PET/CT

INTERVENTIONS:
Diagnostic Test: [18F]MISO-PET/CT — 18F]MISO-PET/CT will be acquired in each patient as the standard of references of tumor hypoxia.

SUMMARY:
Tumor hypoxia is one of the physiological factors for treatment resistance and likely contributes to poor overall survival among patients with head and neck cancer (HNC). Identifying hypoxic features of HNC may allow the personalizing treatment plan. The investigators propose multiparametric Hypoxia MR (HMR) imaging using diffusion, perfusion, and oxygenation as non-invasive, in-vivo imaging components of a hypoxia phenotype. Assessing the hypoxia phenotypes' expression will be critically important for characterizing and predicting CRT response among patients with advanced HNC.

A prospective cohort study will be conducted used multiparametric MR (MPMR) imaging correlated with treatment response assessed by 3 months fluorodeoxyglucose-positron emission tomography (FDG-PET). The image analysis approach will be developed to incorporate FDG-PET and quantitative MRI characteristics of tumor (ADC, oxygen-enhanced T1 and T2* maps, and volume transfer constant (Ktrans) to facilitate 3D visualization of multiparametric information. This proposed study's overarching goal is to develop and validate multiparametric HMR imaging using 18F - (fluoromisonidazole) FMISO-PET and immunohistochemistry (IHC) as the standard of references.

DETAILED DESCRIPTION:
The objectives of this feasibility study are; 1) To obtain pilot data for a full-scale study and measure the distribution of parameters of the hypoxia MR (perfusion, diffusion, oxygenation, and acidosis) imaging, 2) To assess association of various hypoxia MR metrics with outcome, response to chemoradiotherapy (CRT) determined by 3 months post CRT FDG-PET/CT. 3) The metrics developed on hypoxia MRI wil be validated against F-18 FMISO-PET/CT and whole specimen IHC (immunohistochemistry). The data obtained from this pilot study will allow us to measure the effect size (difference in hypoxia MR metrics between responder and non-responder) for a larger, full-scale diagnostic study in the future, as well as to determine which hypoxia MR parameters have a strong association with desired outcome (response to CRT) in the future study.

The long-term objective of this research is to evaluate hypoxia MR phenotype that can be incorporated into treatment planning for IMRT (intensity-modulated radiotherapy), identify subregions of tumor hypoxia, and predict response to chemoradiotherapy (CRT) in newly diagnosed head and neck squamous cell carcinoma. The investigators will develop hypoxia MRI using a widely available MRI platform that allows broad patients access to novel hypoxia MRI. The investigators will evaluate the accuracy of the prediction of response to CRT using quantitative variables derived from hypoxia MR at the baseline as well as early interval changes between the baseline and 2 weeks of intra-treatment MR scans. Response to CRT will be determined by 3 months post-treatment FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HNSCC (head and neck squamous cell carcinoma) by biopsy or fine needle aspiration originating from the oral cavity, larynx, hypopharynx, nasopharynx, and oropharynx
* Patients are scheduled to undergo chemoradiotherapy or surgery
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Pregnant patients
* Patients with claustrophobia
* Patients with pacemaker, spinal stimulator, or cochlear implant that are not MR compatible or any other metallic objects in the body
* Patients who had been treated for HNC, either surgery, radiation therapy, or chemotherapy
* Patients with thyroid, skin, sinonasal, and salivary gland cancer.
* Abnormal kidney function defined as estimated glomerular filtration rate (eGRF) < 30 mL/min/1.73 m2
* Patients with uncontrolled diabetes
* Patients who obtained outside FDG-PET/CT prior to initial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with newly diagnosed advanced-stage HNC with a primary tumor larger than 3 cm that are treated with CRT (chemoradiotherapy)
  2. Patients with newly diagnosed localized HNC that are primarily treated with surgical resection for whole specimen IHC
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The correlation of hypoxia volume between hypoxia MR and F18-FMISO PET | 1 year
  the correlation of the percentages of hypoxia volume on hypoxia MR and F18-FMISO PET as the standard references

SECONDARY OUTCOMES:
The correlation of hypoxia volume between hypoxia MR and IHC with hypoxia biomarkers | 1 year
  Percent volume of the hypoxic subregion measured on both hypoxia MR and IHC
Response to chemoradiotherapy | 1 year
  Correlation with hypoxia phenotype identified on hypoxia MR with response to chemoradiotherapy determined by pre and 3 month post treatment FDG-PET/CT as the standard clinical practice. Those patients with equivocal FDG-PET/CT will be followed clinically and conventional CT or MR imaging up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimi Anzai, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roberts J, Kim SE, Kholmovski EG, Hitchcock Y, Richards TJ, Anzai Y. The arterial input function: Spatial dependence within the imaging volume and its influence on 3D quantitative dynamic contrast-enhanced MRI for head and neck cancer. Magn Reson Imaging. 2023 Sep;101:40-46. doi: 10.1016/j.mri.2023.03.016. Epub 2023 Apr 7. PMID 37030177